CLINICAL TRIAL: NCT00602264
Title: Adipocytokine and Ghrelin Concentrations in Different Stages of Anorexia Nervosa
Brief Title: Adipokines and Ghrelin Concentrations in Different Stages of Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Basak Yucel, Istanbul University Istanbul Medical Faculty Department of Psychiatrics
Other Study IDs: 503/5052006; 2005/1795
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Anorexia Nervosa; Adipokines
Keywords: Anorexia nervosa; Adipokines; Ghrelin; Fat mass
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Treatment-naïve patients with a recent diagnosis of anorexia nervosa
- 2: The weight recovered subgroup of group 1
- 3: Recovered patients with a previous history of anorexia nervosa but normal menstrual cycles and body weight at the present time
- 4: Control group

SUMMARY:
The aim of this study is to determine serum concentrations of adiponectin (ApN), leptin and ghrelin in different stages of anorectic patients and to evaluate their relationships between biochemical, hormonal and anthropometric parameters.

DETAILED DESCRIPTION:
Objective: The aim of this study is to determine serum concentrations of adiponectin (ApN), leptin and ghrelin in different stages of anorectic patients and to evaluate their relationships between biochemical, hormonal and anthropometric parameters.

Design: The study group is composed of four groups. Group1: Treatment-naïve patients with a recent diagnosis of AN (n:19), Group 2: The weight recovered (10 % increase in body weight compared with baseline weight) subgroup of group 1 at the end of a mean 117.72±98.14 days of follow-up (n: 12), Group 3: Recovered patients with a previous history of AN but normal menstrual cycles and body weight at the present time (n:10), Group 4: Control group: constitutionally thin healthy young women with normal menstrual cycles (n:10). Venous blood was obtained for measurements of biochemical parameters, ApN, leptin and ghrelin and body composition was determined by bioimpedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anorexia nervosa for Group 1-3
* Constitutionally thin healthy subjects for Group 4

Exclusion Criteria:

* Medical or psychiatric diagnosis other than anorexia nervosa,
* History of gastrointestinal disease for Group 1-3
* History of eating disorder or gastrointestinal or psychiatric disease for control group

Ages: 16 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with anorexia nervosa and constitutionally thin healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Kubat Uzum, M.D, Study Director — Istanbul University Istanbul Medical Faculty Department of Endocrinology and Metabolism; Basak Yucel, Professor, Principal Investigator — Istanbul University Istanbul Medical Faculty Department of Psychiatrics; Beyhan Omer, Professor, Study Chair — Istanbul University Istanbul Medical Faculty Department of Biochemistry; Nese Colak Ozbey, Professor, Study Director — Istanbul University Istanbul Medical Faculty Department of Endocrinology and Metabolism
Locations (1):
- Istanbul Univetsity, Istanbul Medical Faculty, Department of Psychiatrics, Istanbul, Turkey (Türkiye)